CLINICAL TRIAL: NCT03149991
Title: A Double-Blind, Placebo-Controlled Study of Brexpiprazole Plus Ketamine in Treatment-Resistant Depression (TRD)
Brief Title: A Study of Brexpiprazole Plus Ketamine in Treatment-Resistant Depression (TRD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Vice Chair, Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KETBREX001
Record Dates: First submitted 2017-02-24; First posted 2017-05-11 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Depression
Keywords: treatment resistant; inadequate response
MeSH Terms: conditions — Depression | interventions — brexpiprazole; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine/Brexpiprazole Arm (Active Comparator): brexpiprazole up to 3 mg/day for four weeks in combination with bi-weekly administration of intranasal ketamine (40 mg) for two weeks, followed by weekly administration of intranasal ketamine (40 mg) for two weeks
  Interventions: Drug: Brexpiprazole; Drug: Ketamine
- Ketamine/Placebo Arm (Placebo Comparator): placebo for four weeks in combination with bi-weekly administration of intranasal ketamine (40 mg) for two weeks, followed by weekly administration of intranasal ketamine (40 mg) for two weeks
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Administration of up to 3mg brexpiprazole
  Other Names: rexulti
  Arms: Ketamine/Brexpiprazole Arm
Drug: Ketamine — administration 6 times over two weeks of inhaled ketamine
  Other Names: Inhaled ketamine
Drug: Placebo — Administration of placebo which matches brexpiprazole in size and number of tablets per dose
  Arms: Ketamine/Placebo Arm

SUMMARY:
This is a multi-site, double-blind, placebo-controlled study of the acute efficacy of brexpiprazole or placebo in combination with intranasal ketamine added to ongoing, stable, and adequate antidepressant therapy (ADT) in the treatment of adults with Major Depressive Disorder with Treatment Resistant Depression.

DETAILED DESCRIPTION:
This is a five-site, double-blind, placebo-controlled study of the acute efficacy of oral brexpiprazole or placebo combined with intranasal ketamine added to ongoing, stable, and adequate antidepressant therapy (ADT) in the treatment of adults with MDD with TRD. Adequate ADT is defined as a therapeutically sufficient dose for a sufficient treatment period, which would be expected to be effective as listed in the MGH ATRQ.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 65 years of age, inclusive, at screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
3. Diagnosed with MDD, single or recurrent, and currently experiencing a major depressive episode (MDE) of at least eight weeks in duration, prior to screening, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). The diagnosis of MDD will be made by a site psychiatrist and supported by the SCID-5. The diagnosis will be confirmed by remote, independent raters from the MGH CTNI (Massachusetts General Hospital Clinical Trials Network and Institute) with a SAFER interview.
4. Has a history of treatment resistant depression (TRD) during the current MDE, as assessed by the investigator and remote centralized rater using the MGH ATRQ. TRD is defined as failure to achieve a satisfactory response (e.g., less than 50% improvement of depression symptoms), as perceived by the participant, to at least 2 "treatment courses" during the current episode of a therapeutic dose of an antidepressant therapy (ADT) of at least 8 weeks duration (including the current ADT). The adequacy of dose and duration of the antidepressant therapy will be determined as per the MGH ATRQ criteria. The TRD status will be confirmed by remote, independent raters from the MGH CTNI who will administer the MGH ATRQ, via teleconference, between the screening visit and the baseline visit. Participants must currently be on a stable (for at least 4 weeks) and adequate (according to the MGH ATRQ) dose of ongoing antidepressant therapy (any antidepressant therapy, with the exception of MAOIs), of which total duration must be at least 8 weeks.
5. Meet the threshold on the total MADRS score of >20 at both the screen visit and the baseline visit (Day -7/-28 and Day 0), and as confirmed by the remote centralized MGH CTNI rater between the screen visit and the baseline visit.
6. In good general health, as ascertained by medical history, physical examination (PE) (including measurement of supine and standing vital signs), clinical laboratory evaluations, and ECG.
7. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   * Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or
   * Childbearing potential, and meets the following criteria:

     * Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.
     * Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at randomization prior to receiving study treatment.
     * Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.
8. Body mass index between 18-35 kg/m2.
9. Concurrent psychotherapy will be allowed if the type (e.g., supportive, cognitive behavioral, insight-oriented, et al.) and frequency (e.g., weekly or monthly) of the therapy has been stable for at least three months prior to screening and if the type and frequency of the therapy is expected to remain stable during the course of the subject's participation in the study.
10. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines or trazodone) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study. Patients can also continue treatment with benzodiazepines used for anxiety if therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

Exclusion Criteria:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female that is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or baseline.
4. History during the current MDE of failure to achieve satisfactory response (e.g., less than 50% improvement of depression symptoms) to >7 treatment courses of a therapeutic dose of an antidepressant therapy of at least 8 weeks duration, according to the MGH ATRQ, as confirmed by the remote, independent MGH CTNI rater.
5. Total MADRS score of <20 at the screen visit or the baseline visit, or as assessed by the remote, independent MGH CTNI rater and reported to the site.
6. Current diagnosis of a substance use disorder (abuse or dependence, as defined by DSM-IV-TR™), with the exception of nicotine dependence, at screening or within 6 months prior to screening.
7. Current Axis I disorder, diagnosed at screening with the use of the Structured Clinical Interview for DSM-5 AXIS I Disorders (SCID-5), that is the principal focus of treatment and MDD the secondary focus of treatment for the past 6 months or more.
8. History of bipolar disorder, schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
9. History of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within 5 years of screening.
10. Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within 6 months prior to screening.
11. In the judgment of the investigator, the subject is considered at significant risk for suicidal behavior during the course of his/her participation in the study.
12. Has failed to respond to ECT during the current depressive episode.
13. Has received VNS at any time prior to screening.
14. Has dementia, delirium, amnestic, or any other cognitive disorder.
15. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results according to the study clinician.
16. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
17. Current episode of:

    * Hypertension, Stage 1 as defined by a systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mHg at the Baseline Visit (Visit 1) within 1.5 hours prior to randomization on two of three measurements (standing and supine) at least 15 minutes apart.
    * Recent myocardial infarction (within one year) or a history of myocardial infarction.
    * Syncopal event within the past year.
    * Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2
    * Angina pectoris.
    * Heart rate <45 or >110 beats per minute at screening or randomization (Baseline Visit).
    * QTcF (Fridericia-corrected) ≥450 msec at screening or randomization (Baseline Visit).
18. Chronic lung disease excluding asthma.
19. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention which, according to the screening clinician, is deemed associated with significant injury to or malfunction of the CNS, or history of significant head trauma within the past 2 years.
20. Presents with any of the following lab abnormalities:

    * Thyroid stimulating hormone (TSH) outside of the normal limits and clinically significant as determined by the investigator. Free thyroxine (T4) levels may be measured if TSH level is high. Subject will be excluded if T4 level is clinically significant.
    * Patients with diabetes mellitus fulfilling any of the following criteria:

      * Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.5% at screening.
      * Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus-related illness in the past 12 weeks.
      * Not under physician care for diabetes mellitus.
      * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.
    * Any other clinically significant abnormal laboratory result (determined as such by the investigator and MGH CTNI medical monitor) at the time of the screening.
21. History of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than 2 months prior to screening. (Subjects on a stable dosage of thyroid replacement medication for at least 2 months or more prior to screening are eligible for enrollment.)
22. History of hyperthyroidism which was treated (medically or surgically) less than 6 months prior to screening.
23. History of positive screening urine test for drugs of abuse at screening: cannabinoids (if the patient has a legitimate medical prescription for cannabis, patient must agree to abstain during the entirety of the study and to have a negative test at baseline), cocaine, amphetamines, barbiturates, opiates (unless use is in accordance with guidance provided in table of allowed and excluded medications).
24. Patients with exclusionary laboratory values (see Table 1), or requiring treatment with exclusionary concomitant medications (see Appendix 1).
25. Patients on exclusionary concomitant psychotropic medications, the half-life of which would not allow sufficient time for patients to have been free of the medication post-taper for five half-lives within the maximum screening period (28 days).
26. Patients with a history of narrow angle glaucoma.
27. Liver or renal Function tests which meet the exclusion criteria in Table 1, or a history of hepatic or renal dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - Pacific Research Partners, LLC, Oakland, California
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Depression Clinical and Research Program, Boston, Massachusetts
  - Nathan Kline Institute for Psychiatric Research, Orangeburg, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Started | 25 | 26
Completed Primary Endpoint (Day 14) | 25 | 24
Exited | 4 | 2
Completed | 21 | 24
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (12.4) | 44.6 (13.9) | 42.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 11 | 14 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 22 | 25 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 21 | 23 | 44
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Clinical Severity at Baseline -SDQ [Mean (Standard Deviation); unit: units on a scale] — Symptoms of Depression Questionnaire (SDQ): This validated self-rating instrument has 44 items on a scale of 1-6, measuring multiple depressive symptom domains and with higher scores indicating worse depression symptoms. Participants reported on their experiences over the past 3 days.
  units on a scale | 3.7 (0.6) | 3.7 (0.5) | 3.7 (0.6)
Clinical Severity at Baseline- MADRS [Mean (Standard Deviation); unit: units on a scale] — Montgomery-Asberg Depression Rating Scale (MADRS): This 10-item clinician-rated instrument measures depression severity with higher scores indicating more severity. Each item can be scored from 0 to 6 for a total score range of 0 to 60. Experiences over the past 3 days were rated.
  units on a scale | 33.8 (4.0) | 34.2 (5.5) | 34.0 (4.8)
Clinical Severity at Baseline- HAM-D6 [Mean (Standard Deviation); unit: units on a scale] — 6-item Hamilton Rating Scale for Depression (HAM-D6): This instrument is completed with a structured interview guide developed per Bech by the clinician based on his/her assessment of the patient's symptoms, with higher scores indicating worse depression symptoms. The score ranges from 0-22. Experiences over the past 3 days were rated.
  units on a scale | 12.0 (2.0) | 11.9 (2.2) | 12.0 (2.1)
Clinical Severity at Baseline- CGI-S [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impressions-Severity (CGI-S): This clinician-rated item assesses the severity of the disorder at the time of assessment, relative to the clinician's experiences with patients with the same diagnosis. It involves a 7-point scale ranging from 1=Normal, not at all ill to 7=Among the most extremely ill patients.
  units on a scale | 5.0 (0.6) | 4.8 (0.7) | 4.9 (0.7)
Clinical Severity at Baseline- CGI-I [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impressions-Improvement (CGI-I) Scale: This clinician-rated item assesses global improvement since beginning of the study on a 7-point scale ranging from 1=very much improved to 7=very much worse.
  units on a scale | 4.2 (0.4) | 4.2 (0.5) | 4.2 (0.4)
Duration of Current Major Depressive Episode [Mean (Standard Deviation); unit: years] | 4.6 (6.1) | 4.3 (7.0) | 4.4 (6.5)
Number of current comorbid psychiatric conditions [Mean (Standard Deviation); unit: Conditions] | 0.1 (0.3) | 0.2 (0.5) | 0.1 (0.4)
Number of comorbid medical conditions [Mean (Standard Deviation); unit: Conditions] | 2.6 (2.0) | 2.5 (1.9) | 2.5 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Symptoms of Depression Questionnaire (SDQ)
Description: Superiority will be demonstrated by a statistically significant greater decrease (p<0.05, 2 sided) on the SDQ total score for participants receiving brexpiprazole versus placebo therapy.
  Symptoms of Depression Questionnaire (SDQ): This validated self-rating instrument has 44 items on a scale of 1-6, measuring multiple depressive symptom domains, with higher scores indicating worse depression symptoms. Participants reported on their experiences over the past three days.
Time Frame: SDQ was assessed on Days 0, 1, 2, 5, 8, 11, 14, 17, 21, 23, 28
Population: A total of 54 people were randomized, but only 51 received the study drug or placebo and were included in outcome analyses. Of these, 49 (96%) completed study assessments for the primary endpoint, and n=45 (88%) completed the study. See participant flow data for more information.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
score on a scale
  SDQ, Day 0 | 3.7 (0.6) | 3.7 (0.5)
  SDQ, Day 1 | 3.5 (0.6) | 3.5 (0.6)
  SDQ, Day 2: number analyzed (Participants) | 23 | 26
  SDQ, Day 2 | 3.5 (0.6) | 3.3 (0.6)
  SDQ, Day 5: number analyzed (Participants) | 23 | 24
  SDQ, Day 5 | 3.4 (0.6) | 3.3 (0.6)
  SDQ, Day 8: number analyzed (Participants) | 25 | 24
  SDQ, Day 8 | 3.3 (0.5) | 3.2 (0.5)
  SDQ, Day 11: number analyzed (Participants) | 24 | 24
  SDQ, Day 11 | 3.1 (0.5) | 3.1 (0.6)
  SDQ, Day 14: number analyzed (Participants) | 25 | 24
  SDQ, Day 14 | 3.0 (0.5) | 3.2 (0.7)
  SDQ, Day 17: number analyzed (Participants) | 23 | 23
  SDQ, Day 17 | 3.1 (0.6) | 3.2 (0.7)
  SDQ, Day 21: number analyzed (Participants) | 24 | 23
  SDQ, Day 21 | 3.0 (0.7) | 3.2 (0.6)
  SDQ, Day 23: number analyzed (Participants) | 22 | 23
  SDQ, Day 23 | 2.8 (0.6) | 3.0 (0.6)
  SDQ, Day 28: number analyzed (Participants) | 23 | 25
  SDQ, Day 28 | 2.9 (0.6) | 3.0 (0.6)
Statistical Analysis 1: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; SDQ total was primary outcome & Day 14 primary endpoint. Change from baseline was calculated for each person at each follow-up. Change score was the dependent variable in a linear fixed effects model, where a (-)number = less severe depression. For group comparison, treatment was coded as 1 & placebo as 0, thus a (-)value means treatment doing better. Fixed effects: group(brex v placebo), day(1-28), site(6 sites). All 2-& 3-way interactions were included, as well as a priori defined covariates; Test type: Superiority — The unstructured covariance matrix structure was used to model nesting of observations within persons. Non-significant site interaction effects were removed one at a time. Least squares means estimates of the linear fixed effects model on SDQ change scores, adjusting for baseline covariates was used to test the primary hypothesis via contrast statements; p = 0.46, Mixed Models Analysis; Because sample sizes per site varied substantially, we used the Kenward-Roger degrees of freedom method; Mean Difference (Final Values) = -0.11, Standard Error of Mean 0.15 — degrees of freedom = 44.5; t=-0.74
Statistical Analysis 2: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; Secondary Aim: To evaluate the short-term effect of brexpiprazole, as measured by the Symptoms of Depression Questionnaire (SDQ), on Day 2. We used the same model as in Aim 1 to test this hypothesis; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 0.22, Standard Error of Mean 0.11 — Degrees of freedom = 41.3; t=2.07
Statistical Analysis 3: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; To evaluate the long-term effect of brexpiprazole as measured by the Symptoms of Depression Questionnaire (SDQ) on Day 28. The same model as was used in Aim 1 was used to test this hypothesis; Test type: Superiority; p = 0.92, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, Standard Error of Mean 0.21 — Degrees of freedom=38.2; t=0.10

2. Secondary Outcome: Long-term Sustained Response, as Measured by Achieving a 50% Reduction on the Montgomery-Asberg Depression Rating Scale (MADRS) on Day 28 (Number and Percentage of Participants Achieving Sustained Response Reported)
Description: The table below compares percentages of participants in each arm who achieved a 50% or greater reduction on the Montgomery-Asberg Depression Rating Scale (MADRS) on Day 28 compared with baseline. This 10- item clinician-rated instrument measures depression severity with higher scores indicating more severity. Each item can be scored from 0 to 6 for a total sore range of 0 to 60. It was administered with a structured interview guide. Experiences over the past 3 days were rated.
Time Frame: MADRS was assessed on Days 0, 2, 3, 8, 11, 14, 17, 21, 23, 28; 50% reduction compared Day 28 to Baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Participants | 10 | 8
Statistical Analysis 1: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; We used a Chi-squared test to assess differences between treatment and control in terms of percent of participants achieving a long-term sustained response, as measured by achieving a 50% or greater reduction on the MADRS on Day 28; Test type: Superiority; p = 0.47, Chi-squared — This p-value was not adjusted, however there were adjustments when using a logistic regression in Statistical Analysis #2; Chi-squared test = 0.51
Statistical Analysis 2: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; Logistic regression was used to assess a difference in 50% reduction on the MADRS on Day 28 between groups; Test type: Superiority; p = 0.35, Regression, Logistic; Adjusted for a priori defined covariates also included in Aim 1; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.52 to 6.44]

3. Secondary Outcome: Efficacy on Secondary Outcome Variables
Description: Montgomery-Asberg Depression Rating Scale (MADRS):This 10-item clinician-rated instrument measures depression severity. Total score range of 0-60 with higher scores indicating more severity.
  6-item Hamilton Rating Scale for Depression (HAM-D6): This instrument is completed with a structured interview guide by the clinician based on his/her assessment of the patient's symptoms, with higher scores indicating worse depression. Scores range from 0-22. Experiences were rated based on the past 3 days.
  Clinical Global Impressions-Severity (CGI-S) and Clinical Global Impressions-Improvement (CGI-I) scales: These clinician-rated scales rate the severity of the disorder and the global improvement since beginning of the study. Further information is in the baseline measures section.
Time Frame: These secondary outcome variables were assessed on Days 0, 1 (except for MADRS this day), 2, 5, 8, 11, 14, 17, 21, 23, 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
score on a scale
  MADRS, Day 0 | 33.84 (4.03) | 34.19 (5.54)
  MADRS, Day 2: number analyzed (Participants) | 23 | 26
  MADRS, Day 2 | 31.87 (5.96) | 28.19 (6.79)
  MADRS, Day 5: number analyzed (Participants) | 24 | 24
  MADRS, Day 5 | 29.46 (7.56) | 27.42 (8.75)
  MADRS, Day 8: number analyzed (Participants) | 25 | 25
  MADRS, Day 8 | 27.64 (7.60) | 24.48 (9.16)
  MADRS, Day 11: number analyzed (Participants) | 24 | 24
  MADRS, Day 11 | 23.63 (8.94) | 21.83 (9.95)
  MADRS, Day 14: number analyzed (Participants) | 25 | 24
  MADRS, Day 14 | 21.28 (9.53) | 22.08 (12.10)
  MADRS, Day 17: number analyzed (Participants) | 24 | 23
  MADRS, Day 17 | 20.92 (10.92) | 23.52 (12.07)
  MADRS, Day 21: number analyzed (Participants) | 24 | 24
  MADRS, Day 21 | 20.5 (12.34) | 23.75 (10.63)
  MADRS, Day 23: number analyzed (Participants) | 22 | 23
  MADRS, Day 23 | 18.36 (11.29) | 23.57 (10.53)
  MADRS, Day 28: number analyzed (Participants) | 23 | 24
  MADRS, Day 28 | 18.39 (11.86) | 22.13 (9.98)
  HAMD6, Day 0: number analyzed (Participants) | 7 | 10
  HAMD6, Day 0 | 11 (3.37) | 11.6 (2.07)
  HAMD6, Day 1 | 10.24 (2.35) | 9.19 (3.09)
  HAMD6, Day 2: number analyzed (Participants) | 23 | 26
  HAMD6, Day 2 | 10.48 (2.45) | 8.62 (3.51)
  HAMD6, Day 5: number analyzed (Participants) | 24 | 24
  HAMD6, Day 5 | 10.08 (2.53) | 9.21 (3.09)
  HAMD6, Day 8: number analyzed (Participants) | 25 | 25
  HAMD6, Day 8 | 9.4 (2.58) | 7.64 (4.13)
  HAMD6, Day 11: number analyzed (Participants) | 24 | 24
  HAMD6, Day 11 | 7.96 (3.03) | 7.71 (4.14)
  HAMD6, Day 14: number analyzed (Participants) | 25 | 24
  HAMD6, Day 14 | 7.36 (3.0) | 7.54 (4.68)
  HAMD6, Day 17: number analyzed (Participants) | 24 | 23
  HAMD6, Day 17 | 6.96 (3.79) | 8.09 (4.33)
  HAMD6, Day 21: number analyzed (Participants) | 24 | 24
  HAMD6, Day 21 | 6.83 (3.82) | 7.83 (4.25)
  HAMD6, Day 23: number analyzed (Participants) | 22 | 23
  HAMD6, Day 23 | 6.68 (3.41) | 7.48 (4.18)
  HAMD6, Day 28: number analyzed (Participants) | 23 | 24
  HAMD6, Day 28 | 6.43 (4.04) | 7.58 (3.69)
  CGI-S, Day 0 | 4.96 (0.61) | 4.77 (0.71)
  CGI-S, Day 1 | 4.56 (0.77) | 4.15 (0.73)
  CGI-S, Day 2: number analyzed (Participants) | 23 | 26
  CGI-S, Day 2 | 4.61 (0.66) | 4.12 (0.59)
  CGI-S, Day 5: number analyzed (Participants) | 24 | 24
  CGI-S, Day 5 | 4.33 (0.92) | 4 (1.02)
  CGI-S, Day 8: number analyzed (Participants) | 24 | 25
  CGI-S, Day 8 | 4.29 (0.95) | 3.68 (1.22)
  CGI-S, Day 11: number analyzed (Participants) | 23 | 24
  CGI-S, Day 11 | 3.78 (1.04) | 3.38 (1.13)
  CGI-S, Day 14: number analyzed (Participants) | 25 | 24
  CGI-S, Day 14 | 3.48 (1.08) | 3.33 (1.24)
  CGI-S, Day 17: number analyzed (Participants) | 24 | 23
  CGI-S, Day 17 | 3.42 (1.32) | 3.48 (1.34)
  CGI-S, Day 21: number analyzed (Participants) | 24 | 24
  CGI-S, Day 21 | 3.46 (1.44) | 3.58 (1.21)
  CGI-S, Day 23: number analyzed (Participants) | 22 | 23
  CGI-S, Day 23 | 3.14 (1.39) | 3.48 (1.27)
  CGI-S, Day 28: number analyzed (Participants) | 23 | 24
  CGI-S, Day 28 | 3.17 (1.56) | 3.46 (1.14)
  CGI-I, Day 0 | 4.16 (0.37) | 4.15 (0.46)
  CGI-I, Day 1 | 3.8 (0.5) | 3.35 (0.85)
  CGI-I, Day 2: number analyzed (Participants) | 23 | 26
  CGI-I, Day 2 | 3.65 (0.78) | 3.42 (0.76)
  CGI-I, Day 5: number analyzed (Participants) | 24 | 24
  CGI-I, Day 5 | 3.5 (0.78) | 3.29 (1.0)
  CGI-I, Day 8: number analyzed (Participants) | 25 | 25
  CGI-I, Day 8 | 3.2 (0.87) | 2.92 (1.0)
  CGI-I, Day 11: number analyzed (Participants) | 23 | 24
  CGI-I, Day 11 | 2.87 (0.92) | 2.7 (0.92)
  CGI-I, Day 14: number analyzed (Participants) | 25 | 24
  CGI-I, Day 14 | 2.8 (0.96) | 2.54 (0.98)
  CGI-I, Day 17: number analyzed (Participants) | 24 | 23
  CGI-I, Day 17 | 2.67 (1.09) | 2.83 (1.19)
  CGI-I, Day 21: number analyzed (Participants) | 24 | 24
  CGI-I, Day 21 | 2.75 (1.29) | 2.83 (1.13)
  CGI-I, Day 23: number analyzed (Participants) | 22 | 23
  CGI-I, Day 23 | 2.41 (1.18) | 2.74 (1.14)
  CGI-I, Day 28: number analyzed (Participants) | 23 | 24
  CGI-I, Day 28 | 2.48 (1.27) | 2.54 (1.18)
Statistical Analysis 1: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the MADRS change scores, reporting here information for Day 2; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.04, Mixed Models Analysis — Because tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = 3.39, Standard Error of Mean 1.59 — degrees of freedom = 41.0, t=2.13
Statistical Analysis 2: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the MADRS change scores, reporting here information for Day 14; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.73, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = -1.03, Standard Error of Mean 2.94 — df = 44.2, t=-0.35
Statistical Analysis 3: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the MADRS change scores, reporting here information for Day 28; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.37, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = -2.86, Standard Error of Mean 3.16 — df =44.8, t=-0.91
Statistical Analysis 4: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the HAMD6 change scores, reporting here information for Day 2; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.06, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = 1.66, Standard Error of Mean 0.85 — degrees of freedom = 40.3, t=1.94
Statistical Analysis 5: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the HAMD6 change scores, reporting here information for Day 14; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.83, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = -0.23, Standard Error of Mean 1.06 — df = 44.2, t=-0.22
Statistical Analysis 6: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the HAMD6 change scores, reporting here information for Day 28; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.52, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = -0.77, Standard Error of Mean 1.20 — df =44.0, t=-0.64
Statistical Analysis 7: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the CGI-S change scores, reporting here information for Day 2; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.11, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = 0.31, Standard Error of Mean 0.19 — df = 31.0, t=1.67
Statistical Analysis 8: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the CGI-S change scores, reporting here information for Day 14; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.98, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Net) = -0.01, Standard Error of Mean 0.36 — df=41.1, t=-0.03
Statistical Analysis 9: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the CGI-S change scores, reporting here information for Day 28; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest; p = 0.45, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = -0.31, Standard Error of Mean 0.41 — df=46.0, t=-0.76
Statistical Analysis 10: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the CGI-I change scores, reporting here information for Day 2; Test type: Superiority — We used contrast tests comparing brexpiprazole and placebo on the a priori specified days of interest. This model contains an interaction effect with site, because the SITE*DRUG effect was significant (p=0.03); p = 0.02, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = 0.69, Standard Error of Mean 0.29 — df=49.2, t=2.39;
Statistical Analysis 11: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the CGI-I change scores, reporting here information for Day 14; Test type: Superiority — [test comment as in outcome 3, analysis 10]; p = 0.07, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = 0.63, Standard Error of Mean 0.34 — df=56.8, t=1.85
Statistical Analysis 12: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; The same model building approach as used for the primary outcome variable was used for the secondary outcome variables. As per the primary outcome variable, the change scores (i.e., compared to baseline) were the dependent variables of interest. For each secondary outcome variable, non-significant site interaction effects were removed one at a time. This analysis is for the CGI-I change scores, reporting here information for Day 28; Test type: Superiority — [test comment as in outcome 3, analysis 10]; p = 0.37, Mixed Models Analysis — Because these tests were conducted for secondary outcomes, p-values were not corrected for multiple testing; Mean Difference (Final Values) = 0.37, Standard Error of Mean 0.41 — df=50.5, t=0.91

4. Secondary Outcome: Safety and Tolerability Outcomes: Number of Participants With Abnormal Vital Signs (Elevated Blood Pressure)
Description: Blood pressure was measured during each administration of ketamine, occurring on days 0, 5, 8, 11, 14, and 21. This vital sign was measured 6 times following the intranasal administration of ketamine: 15 minutes post dose, 30 minutes post dose, 45 minutes post dose, 1 hour post dose, 90 minutes post dose, and 2 hours post dose. Average blood pressure per group was assessed. Medical staff monitoring the ketamine administration were prepared to treat increases in blood pressure greater than 180/110 mm Hg or follow their institutional guidelines if more conservative, if these elevations did not resolve spontaneously within a short time period. Data presented are number of participants with elevated blood pressure at any of the listed time points.
Time Frame: Blood pressure was measured during each administration of ketamine, occurring on days 0, 5, 8, 11, 14, and 21. This vital sign was measured 6 times following the intranasal administration of ketamine: 15 minutes post dose, 30 minutes post dose, 45 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Participants | 1 | 0

5. Secondary Outcome: Safety and Tolerability Outcomes: Number of Participants With Abnormal Vital Signs (Elevated Heart Rate)
Description: Heart rate was measured during each administration of ketamine, occurring on days 0, 5, 8, 11, 14, and 21. This vital sign was measured 6 times following the intranasal administration of ketamine: 15 minutes post dose, 30 minutes post dose, 45 minutes post dose, 1 hour post dose, 90 minutes post dose, and 2 hours post dose. Average heart rate per group was assessed. Medical staff monitoring the ketamine administration were prepared to treat heart rate greater than 110 bpm, or follow their institutional guidelines if more conservative, if these elevations did not resolve spontaneously within a short time period. Data presented are number of participants with elevated heart rate at any of the listed time points.
Time Frame: Heart rate was measured during each administration of ketamine, occurring on days 0, 5, 8, 11, 14, and 21.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Participants | 1 | 1

6. Secondary Outcome: Safety and Tolerability Outcomes: 12-lead Electrocardiogram (ECG) - Total Number of Abnormal ECGs
Description: Electrocardiograms (ECGs) were conducted at baseline, and follow-up visits conducted 5, 8, 11, 14, and 21 days after baseline. Any found to be abnormal were evaluated by a clinician as to the clinical significance of the ECG abnormality.
Time Frame: ECGs were conducted at baseline and 5, 8, 11, 14, and 21 days after baseline
Population: as for outcome 1
Measure: Number; unit: Number of abnormal ECGs
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Number of abnormal ECGs | 60 | 56

7. Secondary Outcome: Safety and Tolerability Outcomes: 12-lead Electrocardiogram (ECG) - Number of Participants With Abnormal ECGs
Description: as for outcome 6
Time Frame: ECGs were conducted at baseline and 5, 8, 11, 14, and 21 days after baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
participants
  # of participants with abnormal ECGs, Baseline | 12 | 9
  # of participants with abnormal ECGs, Day 5: number analyzed (Participants) | 24 | 24
  # of participants with abnormal ECGs, Day 5 | 9 | 9
  # of participants with abnormal ECGs, Day 8: number analyzed (Participants) | 25 | 25
  # of participants with abnormal ECGs, Day 8 | 11 | 12
  # of participants with abnormal ECGs, Day 11: number analyzed (Participants) | 23 | 24
  # of participants with abnormal ECGs, Day 11 | 10 | 10
  # of participants with abnormal ECGs, Day 14: number analyzed (Participants) | 25 | 24
  # of participants with abnormal ECGs, Day 14 | 10 | 7
  # of participants with abnormal ECGs, Day 21: number analyzed (Participants) | 24 | 24
  # of participants with abnormal ECGs, Day 21 | 8 | 9
Statistical Analysis 1: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to assess group differences (drug vs. placebo) in terms of number of abnormal ECGs out of total ECGs assessed; Test type: Equivalence — The hypothesis was that there would be no group differences in terms of occurrence of abnormal ECGs; p = 0.60, Chi-squared; Chi-squared test = 0.28
Statistical Analysis 2: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to assess for group differences (drug vs. placebo) in number/percentage of people with an abnormal ECG at baseline; Test type: Equivalence — The hypothesis was that there would be no group differences in number/percentage of people with an abnormal ECG at baseline; p = 0.33, Chi-squared; Chi-squared test = 0.94
Statistical Analysis 3: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to assess for group differences (drug vs. placebo) in number/percentage of people with an abnormal ECG at Visit 4; Test type: Equivalence — The hypothesis was that there would be no group differences in number/percentage of people with an abnormal ECG at Visit 4; p = 1.00, Chi-squared; Chi-squared test = 0.00
Statistical Analysis 4: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to assess for group differences (drug vs. placebo) in number/percentage of people with an abnormal ECG at Visit 5; Test type: Equivalence — The hypothesis was that there would be no group differences in number/percentage of people with an abnormal ECG at Visit 5; p = 0.78, Chi-squared; Chi-squared test = 0.08
Statistical Analysis 5: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to assess for group differences (drug vs. placebo) in number/percentage of people with an abnormal ECG at Visit 6; Test type: Equivalence — The hypothesis was that there would be no group differences in number/percentage of people with an abnormal ECG at Visit 6; p = 0.90, Chi-squared; Chi-squared test = 0.02
Statistical Analysis 6: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to assess for group differences (drug vs. placebo) in number/percentage of people with an abnormal ECG at Visit 7; Test type: Equivalence — The hypothesis was that there would be no group differences in number/percentage of people with an abnormal ECG at Visit 7; p = 0.43, Chi-squared; Chi-squared test = 0.63
Statistical Analysis 7: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to assess for group differences (drug vs. placebo) in number/percentage of people with an abnormal ECG at Visit 9; Test type: Equivalence — The hypothesis was that there would be no group differences in number/percentage of people with an abnormal ECG at Visit 9; p = 0.76, Chi-squared; Chi-squared test = 0.09

8. Secondary Outcome: Safety and Tolerability Outcomes: Number of Participants With Abnormal Laboratory Test Results
Description: Chemistry and CBC laboratory tests were obtained during the screening visit and on Day 14 and 28 follow-ups. If a test result was abnormal (i.e., outside of the site-specific pre-specified range of expected values), it was evaluated by a clinician as to its clinical significance.
Time Frame: Chemistry and CBC laboratory tests were obtained during screening and on Day 14 and 28 follow-ups
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Participants
  Abnormal lab results at Screening | 1 | 2
  Abnormal lab results at Day 14 | 1 | 0
  Abnormal lab results at Day 28 | 1 | 0

9. Secondary Outcome: Safety and Tolerability Outcomes: Treatment-emergent Adverse Events (Number of Participants Reporting)
Description: Adverse events were recorded on a rolling basis from screening until the last day of the study (i.e., Day 28). For patients who reported any AEs, the average number of AEs per person per group were recorded. Site investigators rated whether AEs were possibly or probably related to treatment.
Time Frame: Adverse events were recorded on a rolling basis from screening through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Participants | 17 | 18
Statistical Analysis 1: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis assessed group differences (drug vs. placebo) in terms of number of participants reporting adverse events; Test type: Equivalence — The hypothesis was that there would be no group differences in number of participants reporting adverse events; p = 0.92, Chi-squared; Chi-squared test = 0.009

10. Secondary Outcome: Safety and Tolerability Outcomes: Treatment-emergent Adverse Events (Average Number Per Person Per Group)
Description: Adverse events were recorded on a rolling basis from screening until the last day of the study (i.e., Day 28). For patients who reported any adverse events, the mean number of adverse events per person per group were calculated and are reported below.
Time Frame: The outcome was recorded on a rolling basis from screening through Day 28
Measure: Mean (Standard Error); unit: Adverse events
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Adverse events | 3.8 (3.1) | 3.6 (3.5)
Statistical Analysis 1: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis assessed group differences (drug vs. placebo) in terms of mean number of adverse events per person, among those who reported any adverse events; Test type: Equivalence — The hypothesis was that there would be no difference between the groups in terms of mean number of adverse events per person, among those who reported any adverse events; p = 0.81, t-test, 2 sided; Mean Difference (Final Values) = 0.24

11. Secondary Outcome: Safety and Tolerability Outcomes: Suicidal Ideation and Behavior
Description: The clinician rated behavioral module of the Concise Health Risk Tracking (CHRT) scale was used at each study visit to identify suicidal ideation and behavior. The first item assesses suicidal ideation. All subsequent items assess suicidal behavior. The below table is for Item 1.
Time Frame: The CHRT was used at each study visit through Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine/Brexpiprazole Arm | Ketamine/Placebo Arm
Number analyzed (Participants) | 25 | 26
Participants
  Suicidal Ideation-Screening | 9 | 4
  Suicidal Ideation-Baseline | 4 | 4
  Suicidal Ideation-Day 1 | 5 | 5
  Suicidal Ideation-Day 2: number analyzed (Participants) | 23 | 26
  Suicidal Ideation-Day 2 | 5 | 2
  Suicidal Ideation-Day 5: number analyzed (Participants) | 24 | 24
  Suicidal Ideation-Day 5 | 5 | 7
  Suicidal Ideation-Day 8: number analyzed (Participants) | 25 | 25
  Suicidal Ideation-Day 8 | 5 | 8
  Suicidal Ideation-Day 11: number analyzed (Participants) | 23 | 24
  Suicidal Ideation-Day 11 | 3 | 3
  Suicidal Ideation-Day 14: number analyzed (Participants) | 25 | 24
  Suicidal Ideation-Day 14 | 5 | 3
  Suicidal Ideation-Day 17: number analyzed (Participants) | 24 | 23
  Suicidal Ideation-Day 17 | 4 | 2
  Suicidal Ideation-Day 21: number analyzed (Participants) | 24 | 24
  Suicidal Ideation-Day 21 | 4 | 3
  Suicidal Ideation-Day 23: number analyzed (Participants) | 22 | 23
  Suicidal Ideation-Day 23 | 2 | 4
  Suicidal Ideation-Day 28: number analyzed (Participants) | 23 | 24
  Suicidal Ideation-Day 28 | 2 | 4
Statistical Analysis 1: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) throughout the trial; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.51, Chi-squared; Chi-squared test = 0.43
Statistical Analysis 2: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) at Screening; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.09, Chi-squared; Chi-squared = 2.85
Statistical Analysis 3: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) at Baseline; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.95, Chi-squared; Chi-squared = 0.004
Statistical Analysis 4: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 1; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.94, Chi-squared; Chi-squared = 0.005
Statistical Analysis 5: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 2; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.16, Chi-squared; Chi-squared = 1.97
Statistical Analysis 6: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 5; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.51, Chi-squared; Chi-squared = 0.44
Statistical Analysis 7: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 8; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.33, Chi-squared; Chi-squared = 0.94
Statistical Analysis 8: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 11; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.96, Chi-squared; Chi-squared = 0.003
Statistical Analysis 9: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 14; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.48, Chi-squared; Chi-squared = 0.50
Statistical Analysis 10: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 17; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.41, Chi-squared; Chi-squared = 0.67
Statistical Analysis 11: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 21; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.68, Chi-squared; Chi-squared = 0.17
Statistical Analysis 12: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 23; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.41, Chi-squared; Chi-squared = 0.67
Statistical Analysis 13: Comparison: Ketamine/Brexpiprazole Arm vs Ketamine/Placebo Arm; This analysis was to compare by group (drug vs. placebo) the occurrence of suicidal ideation (endorsement of item 1 on the CHRT) on Day 28; Test type: Equivalence — The hypothesis was that there would be no group differences in occurrence of suicidal ideation; p = 0.41, Chi-squared; Chi-squared = 0.67

ADVERSE EVENTS:
Time Frame: Adverse events were recorded on a rolling basis from screening until the last day of the study (i.e., Day 28).
Groups:
- Brexpiprazole: Brexpiprazole combined with intranasal ketamine
- Placebo: Placebo combined with intranasal ketamine
Arm/Group | Brexpiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 17/25 | 18/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=25) | Placebo (N=26)
Dizziness (Ear and labyrinth disorders) | 4 | 7
Headache (General disorders) | 2 | 6
Alteration in Taste (Nervous system disorders) | 4 | 2
Dissociation/Detachment (Psychiatric disorders) | 2 | 3
Insomnia/Sleep disturbance (General disorders) | 2 | 3
Restlessness/Akathisia (Nervous system disorders) | 3 | 1
Sedation (General disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Euphoria (Psychiatric disorders) | 1 | 1
Gastric Distress (Gastrointestinal disorders) | 2 | 0
Irregular/Early Menses (Reproductive system and breast disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Bi-lateral hand pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurred vision (Eye disorders) | 0 | 1
Bruxism (General disorders) | 1 | 0
Diplopia (Nervous system disorders) | 0 | 1
Dry mouth (General disorders) | 0 | 1
Elevated alt (Hepatobiliary disorders) | 1 | 0
Hot flashes (Reproductive system and breast disorders) | 1 | 0
Increased salivation post dose (General disorders) | 1 | 0
Increased appetite (Gastrointestinal disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Lethargy (General disorders) | 1 | 0
Light headedness (General disorders) | 1 | 0
Lower extremity edema, bilateral (General disorders) | 0 | 1
Muscle aches (Musculoskeletal and connective tissue disorders) | 0 | 1
Panic episode (Psychiatric disorders) | 1 | 0
Restless legs (Nervous system disorders) | 0 | 1
Shakiness (General disorders) | 1 | 0
Tachycardia (General disorders) | 0 | 1
Tinnitus (Nervous system disorders) | 0 | 1
Twitching of left side lower lip (Nervous system disorders) | 1 | 0
Unsteadiness of gait (Nervous system disorders) | 1 | 0
Urinary hesitancy (Renal and urinary disorders) | 0 | 1
Vivid dreams (Psychiatric disorders) | 0 | 1
Weight gain (Metabolism and nutrition disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03149991/Prot_SAP_000.pdf